CLINICAL TRIAL: NCT06159101
Title: A Randomized, Intravenous Single-Dose, Parallel, Phase I Clinical Study to Compare the Pharmacokinetic Characteristics, Safety, and Immunogenicity of HLX13 and YERVOY® (US-, EU-, and CN-Sourced) in Healthy Chinese Male Subjects
Brief Title: A Study to Compare the PK , Safety, Tolerability, and Immunogenicity of HLX13 With YERVOY in Male Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX13-001
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Healthy Male Volunteers
Keywords: CTLA-4
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Dependent, 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HLX13 group (Experimental): Recombinant anti-CTLA-4 fully human monoclonal antibody injection developed by Shanghai Henlius Biotech, Inc.
  Interventions: Drug: HLX13
- CN-sourced ipilimumab group (Active Comparator): CN-sourced ipilimumab
  Interventions: Drug: CN-sourced ipilimumab
- EU-sourced ipilimumab group (Active Comparator): EU-sourced ipilimumab
  Interventions: Drug: EU-sourced ipilimumab group
- US-sourced ipilimumab group (Active Comparator): US-sourced ipilimumab
  Interventions: Drug: US-sourced ipilimumab group

INTERVENTIONS:
Drug: HLX13 — A single dose (0.3 mg/kg) of HLX13 via intravenous infusion.
  Arms: HLX13 group
Drug: CN-sourced ipilimumab — A single dose (0.3 mg/kg) of CN-sourced ipilimumab via intravenous infusion.
  Arms: CN-sourced ipilimumab group
Drug: EU-sourced ipilimumab group — A single dose (0.3 mg/kg) of EU-sourced ipilimumab via intravenous infusion.
  Arms: EU-sourced ipilimumab group
Drug: US-sourced ipilimumab group — A single dose (0.3 mg/kg) of US-sourced ipilimumab via intravenous infusion.
  Arms: US-sourced ipilimumab group

SUMMARY:
Phase I Study to Compare the Pharmacokinetic Characteristics, Safety, Tolerability, and Immunogenicity (Randomized, Double-blind, Parallel Controlled) of HLX13 with YERVOY® Injection in Healthy Chinese Male Subjects

DETAILED DESCRIPTION:
This is a randomized, intravenous single-dose, parallel study to compare the PK characteristics of HLX13 and YERVOY® (US-, EU-, and CN-sourced) and evaluate their safety, tolerability, and immunogenicity in healthy Chinese male subjects.

This study is divided into two parts. Part I is an open-label, randomized, single-dose, parallel study to compare the PK parameters of HLX13 with those of EU-sourced YERVOY® in healthy Chinese male subjects after a single intravenous infusion and provide supporting data for the design of Part II. This part of the study consists of two groups.

Part II is a double-blind, randomized, single-dose, parallel study to evaluate the PK similarity of HLX 13 and YERVOY® (US-, EU-, and CN-sourced) in healthy Chinese male subjects. This part of the study consists of four groups.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent form.
2. Healthy Chinese males (no significant clinical abnormalities in medical history, physical examination, vital signs, chest X-ray, 12-lead ECG, and laboratory examinations).
3. Age ≥ 18 and ≤ 60 years old.
4. Body mass index (BMI) ≥ 18.5 and ≤ 28 kg/m2.
5. Left ventricular ejection fraction (LVEF) > 50%, as measured by echocardiography within 14 days before randomization.
6. Subjects either agree that they and their spouse/partner will take reliable contraceptive measures within 3 months after the end of drug infusion or be infertile.

Exclusion Criteria:

1. History of any severe hematological or renal, endocrinic, respiratory, gastrointestinal, cardiovascular, hepatic, neuropsychiatric, or neurological diseases or tumors.
2. Use of a monoclonal antibody or any biological product within 6 months prior to the study treatment.
3. History of allergy or anaphylaxis, including that due to any drug or drug excipients in clinical studies.
4. Use of prescription/over-the-counter drugs or traditional Chinese medicines (except vitamins, mineral supplements, and health products) within 28 days prior to the study treatment.
5. History of blood donation within 3 months prior to the study treatment.
6. Participation in another clinical study and use of a clinical investigational drug or reference product within 3 months prior to the study treatment, or planning to participate in another drug clinical trial during the study period.
7. Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, or Treponema pallidum antibody.
8. History of drug abuse, or positive urine drug screen during the screening period.
9. Have undergone surgery within 3 months before screening or plan to undergo surgery during the study period; have undergone surgery that will affect drug absorption, distribution, metabolism, and excretion.
10. Have been vaccinated within 28 days prior to screening or plan to be vaccinated during the study.
11. Intolerant to venipuncture or with a history of needle or blood phobia.
12. People on special diets who reject the arranged meals.
13. Smoking more than 5 cigarettes per day within 3 months before screening or cannot stop using any tobacco products during the study.
14. An average daily alcohol intake of more than 15 g (equivalent to 450 mL beer or 150 mL wine or 50 mL low-alcohol liquor) within 1 month prior to screening; or a positive blood alcohol test at screening; or unwilling or unable to abstain from alcohol during the study.
15. Failure to comply with protocol requirements and instructions, protocol restrictions, etc., as judged by the investigator; uncooperative or unable to return to the study site for follow-up visits or complete the entire clinical study process, etc.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 304 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-05-28 (Estimated); Study Completion 2024-05-28 (Estimated)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve from time 0 to infinity (AUC0-inf) | Up to Day 90
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Maximum (peak) serum drug concentration (Cmax) | Up to Day 90
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan

SECONDARY OUTCOMES:
Area under the serum concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC0-t) | Up to Day 90
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Percentage of area under the serum concentration-time curve extrapolated to infinity (%AUCex) | Up to Day 90
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Time to reach maximum (peak) serum drug concentration (Tmax) | Up to Day 90
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Elimination half life (t1/2) | Up to Day 90
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Total clearance (CL) | Up to Day 90
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Apparent volume of distribution during terminal phase (Vz) | Up to Day 90
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Mean residence time (MRT) | Up to Day 90
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan

OTHER OUTCOMES:
Adverse events (AEs), serious adverse events (SAEs), | Up to Day 90
Incidence of anti-drug antibodies (ADAs) | Up to Day 90
Incidence of neutralizing antibodies (NAbs). | Up to Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Hu Wei, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Hospital of Anhui Medical University, Anhui, Anhui, China

IPD SHARING:
Plan to Share IPD: No